CLINICAL TRIAL: NCT00324298
Title: A Randomized Phase III Toxicity Study of Day 2, 3, 8, 15 Short (30 Minute) Versus Day 1, 2, 3 Long (72 Hours) Infusion Bleomycin for Patients With IGCCCG Good Prognosis Germ Cell Tumors, TE3
Brief Title: Bleomycin, Etoposide, and Cisplatin in Treating Patients With Metastatic Germ Cell Cancer of the Testicles
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: BARTS-TE3; CDR0000472976 (Registry Identifier: PDQ (Physician Data Query)); EU-20608; ISRCTN08648791
Record Dates: First submitted 2006-05-10; First posted 2006-05-11 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2007-01

CONDITIONS: Drug/Agent Toxicity by Tissue/Organ; Testicular Germ Cell Tumor
Keywords: drug/agent toxicity by tissue/organ; stage III malignant testicular germ cell tumor
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Testicular Germ Cell Tumor; Testicular Neoplasms | interventions — Bleomycin; Cisplatin; Etoposide

INTERVENTIONS:
Biological: bleomycin sulfate
Drug: cisplatin
Drug: etoposide
Procedure: management of therapy complications

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as bleomycin, etoposide, and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. It is not yet known which schedule of bleomycin is more effective when given together with etoposide and cisplatin in treating metastatic germ cell cancer of the testicles.

PURPOSE: This randomized phase III trial is studying two different schedules of bleomycin to compare how well they work when given together with etoposide and cisplatin in treating patients with metastatic germ cell cancer of the testicles.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine if long-infusion schedule of bleomycin is less toxic to the lungs than short-infusion schedule of bleomycin in patients who are undergoing combination chemotherapy comprising bleomycin, etoposide, and cisplatin for good-prognosis, metastatic germ cell cancer of the testes.
* Determine if early lung function tests are a predictor for late toxicity.
* Determine if any indication of enhanced response to the long-infusion schedule justifies a large-scale phase III evaluation.
* Validate the O'Sullivan et al prognostic scoring system for bleomycin toxicity.

Secondary

* Determine response to treatment.
* Determine progression-free survival and overall survival of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to age (≤ 30 years vs > 30 years), current smoker or has smoked within the past 1 year (yes vs no), and creatinine clearance (≤ 80 mL/min vs > 80 mL/min). Patients are randomized to 1 of 2 treatment arms.

* Arm I (short-infusion schedule of bleomycin): Patients receive etoposide IV over 2 hours on days 1-3, cisplatin IV over 4 hours on days 1 and 2, and bleomycin IV over 30 minutes on days 2, 8, and 15.
* Arm II (long-infusion schedule of bleomycin): Patients receive etoposide and cisplatin as in arm I. Patients also receive bleomycin IV continuously over 72 hours on days 1-3.

In both arms, treatment repeats every 3 weeks for up to 3 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 4 weeks and then every 3 months for 24 months.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 210 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of metastatic germ cell cancer of the testes

  * Good-prognosis disease
* Eligible for treatment with bleomycin, etoposide, and cisplatin

PATIENT CHARACTERISTICS:

* Creatinine clearance ≥ 60 mL/min
* No other prior or concurrent malignancy except basal cell skin cancer
* No other major systemic illness
* No impaired respiratory function, including any of the following:

  * Shortness of breath on minimal exertion
  * Hypoxia at rest
* Carbon monoxide transfer, total lung capacity, and FEV_1 > 60% of predicted

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or radiotherapy

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 210 (Estimated)
Dates: Start 2003-07; Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Pulmonary toxicity

SECONDARY OUTCOMES:
Response to treatment
Progression-free survival
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Shamash, MD, FRCP, Study Chair — St. Bartholomew's Hospital
Locations (10):
- United Kingdom (10):
  - Basildon University Hospital, Basildon, England
  - Addenbrooke's Hospital, Cambridge, England
  - Essex County Hospital, Colchester, England
  - Ipswich Hospital, Ipswich, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Saint Bartholomew's Hospital, London, England
  - University College of London Hospitals, London, England
  - Norfolk and Norwich University Hospital, Norwich, England
  - Royal Marsden - Surrey, Sutton, England
  - Southend University Hospital NHS Foundation Trust, Westcliff-on-Sea, England